CLINICAL TRIAL: NCT05347199
Title: Effects of a Single Dose of Amisulpride on Functional Brain Changes During Reward- and Motivation-related Processing
Brief Title: Effects of a Single Dose of Amisulpride on Functional Brain Changes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Simone Grimm (Other)
Collaborators: Charité Research Organisation GmbH (Other); Boehringer Ingelheim (Industry)
Responsible Party: Sponsor-Investigator, Simone Grimm, Prof. Dr. habil., Medical School Berlin
Organization: Medical School Berlin (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MSB-C002
Record Dates: First submitted 2022-04-12; First posted 2022-04-26 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; Amisulpride; Functional Brain Changes; BOLD responses
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Amisulpride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Healthy Volunteers Placebo (Placebo Comparator): placebo pill at two time points
  Interventions: Drug: Placebo
- Healthy Volunteers Amisulpride (Active Comparator): amisulpride pill at two time points
  Interventions: Drug: Amisulpride Pill
- MDD Patients Placebo (Active Comparator): placebo pill at two time points
  Interventions: Drug: Placebo
- MDD Patients Amisulpride (Experimental): amisulpride pill at two time points
  Interventions: Drug: Amisulpride Pill

INTERVENTIONS:
Drug: Amisulpride Pill — Two single low doses amisulpride (100 mg); orally
  Arms: Healthy Volunteers Amisulpride; MDD Patients Amisulpride
Drug: Placebo — two doses, orally
  Arms: Healthy Volunteers Placebo; MDD Patients Placebo

SUMMARY:
This study is designed to investigate effects of a single dose of amisulpride on functional brain changes during reward- and motivation-related processing and at rest in healthy volunteers (HV) and in patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
Double blind, placebo-controlled, randomized, single dose, parallel-group design The study is designed to investigate effects of a single dose of amisulpride on functional brain changes during reward- and motivation-related processing and at rest. Measurement of functional brain changes will occur after a single dose of amisulpride or placebo in HV and patients with MDD. It is hypothesized that functional brain changes previously linked to reward- and motivation-related processing require dopaminergic signaling and are diminished in MDD compared to HV. In MDD, but not in HV, treatment with a single low dose (100 mg) amisulpride should increase brain activation associated with reward- and motivation-related processing. To test these hypotheses, we will implement a randomized, placebo-controlled, parallel- group design with 4 treatment arms (MDD/placebo, MDD/amisulpride, HV/placebo and HV/ amisulpride). All subjects will undergo MRI scanning sessions at Visit 3 and Visit 4. Treatment with amisulpride or matching placebo will occur 3.5 to 4 hours before the start of each scanning session. Time of treatment will be standardized across subjects.

At Visit 3 and Visit 4, blood samples will be taken 30 minutes pre-dose, and 1 hour, 3.5 to 4 hours, and 4.5 to 5 hours after oral drug administration to determine target plasma levels of amisulpride.

The study is composed of 4 outpatient visits: Screening, baseline and 2 scanning sessions.

ELIGIBILITY:
MDD Patients:

Inclusion:

* Male and female patients with MDD; aged 18 to 45 years
* Montgomery-Åsberg Depression Rating Scale (MADRS) score > 7 and <26 at screening.

Exclusion:

* Meeting diagnostic criteria for any major psychiatric disorder (other than MDD), as determined by DSM-5 at screening.
* Having received prescribed medication (including antidepressants (AD)) within 14 days or fluoxetine within 90 days prior to Visit 3 (apart from the contraceptive pill).
* Having received psychotherapy within 14 days prior to Visit 3.
* Positive severe acute respiratory syndrome coronavirus type 2 (SARS-CoV-2) test.

Healthy Volunteers:

Inclusion:

* Healthy
* aged 18 to 45 years

Exclusion:

* Meeting diagnostic criteria for any major psychiatric disorder.
* A history of psychiatric or neurologic disorders.
* Having received prescribed medication within 14 days prior to Visit 3 (apart from the contraceptive pill).
* Positive SARS-CoV-2 test.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 127 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2023-09-18 (Actual); Study Completion 2023-09-25 (Actual)

PRIMARY OUTCOMES:
BOLD fMRI parameter estimates | during MID task at treatment day 1
  Blood oxygen level dependent (BOLD) fMRI parameter estimates (ß-weights within the GLM analysis) will be extracted from task-related regions of interest (average %BOLD signal change and 90th percentile thereof within ROIs) under the following task-specific contrasts:
  Monetary Incentive Delay (MID) task:
  Contrast of 'High-gain'vs. 'No-gain' condition during the task CUE period ROIs ventral striatum (including nucleus accumbens)

OTHER OUTCOMES:
Exploratory endpoint: average %BOLD signal change and 90th percentile thereof within ROIs during SID | during SID task at treatment day 2
  Blood oxygen level dependent (BOLD) fMRI parameter estimates (ß-weights within the GLM analysis) will be extracted from task-related regions of interest (average %BOLD signal change and 90th percentile thereof within ROIs) under the following task-specific contrasts:
  Social Incentive Delay (SID) task:
  Contrast of 'High-gain' vs. 'No-gain' condition during the task CUE period ROIs: ventral striatum (including nucelues accumbens), ventral tegmental area, dorsal anterior cingulate cortex, insula, ventromedial prefrontal cortex/ orbitofrontal cortex and ventral pallidum
Exploratory endpoint: average %BOLD signal change and 90th percentile thereof within ROIs during intstrumental learning task | during instrumental learning task at treatment day 1
  Blood oxygen level dependent (BOLD) fMRI parameter estimates (ß-weights within the GLM analysis) will be extracted from task-related regions of interest (average %BOLD signal change and 90th percentile thereof within ROIs) under the following task-specific contrasts:
  Instrumental Learning task:
  Contrast of the Gain-cue vs. neutral cue conditions during the task cue and feedback periods
  ROIs:
  ventral striatum (including nucelues accumbens), ventral tegmental area, dorsal anterior cingulate cortex, insula, ventromedial prefrontal cortex/ orbitofrontal cortex and ventral pallidum
Exploratory endpoint: average %BOLD signal change and 90th percentile thereof within ROIs during effort-based decision making task | during effort-based decision making task at treatment day 2
  Blood oxygen level dependent (BOLD) fMRI parameter estimates (ß-weights within the GLM analysis) will be extracted from task-related regions of interest (average %BOLD signal change and 90th percentile thereof within ROIs) under the following task-specific contrasts:
  Effort-based Decision Making task:
  Contrast of the High reward vs. Low reward conditions during the task CUE2 period Contrast of the High effort vs. Low effort conditions during the task CUE2 period
  ROIs:
  ventral striatum (including nucelues accumbens), ventral tegmental area, dorsal anterior cingulate cortex, insula, ventromedial prefrontal cortex/ orbitofrontal cortex and ventral pallidum
Exploratory endpoint: reaction times in ms | during all tasks at treatment day 1 and day 2
  Reaction times in ms extracted from the in- scanner protocol log files
Exploratory endpoint: response accuracy in percent | during all tasks at treatment day 1 and day 2
  Estimates of response accuracy extracted from the in- scanner protocol log files
Exploratory endpoint:average %BOLD signal change and 90th percentile thereof within ROIs during resting state | during resting state at treatment day 1
  Blood oxygen level dependent (BOLD) fMRI signal magnitude and BOLD signal standard deviation during Resting State within the following a-priori defined regions:
  Default Mode Network (posterior cingulate, vmPFC and medial temporal lobe), Central Executive Network (dorsolateral prefrontal cortex, premotor cortex, precuneus), and Salience Network Network (amygdala, insula and dorsal anterior cingulate)
Exploratory endpoint: Arterial Spin Labeling (ASL) | during asl at treatment day 1
  Changes in relative and absolute cerebral blood flow measured through Arterial Spin Labelling MR in whole brain and in the following brain regions:
  (bilateral): ventral striatum, ventromedial prefrontal cortex/ orbitofrontal cortex, ventral tegmental area, dorsal anterior cingulate cortex, insula, and ventral pallidum after amisulpride administration
Exploratory endpoint (Correlation between BOLD signal and self-reported anhedonia ) | treatment day 1 and treatment day 2
  Correlation between magnitude of BOLD signal during reward-and motivation-related processing and self-reported anhedonia after amisulpride administration as compared to placebo in MDD patients relative to HV
Exploratory endpoint (Correlation between BOLD signal and behavioral measures) | treatment day 1 and treatment day 2
  Correlation between magnitude of BOLD signal during reward-and motivation-related processing and behavioral measures after amisulpride administration as compared to placebo in MDD patients relative to HV
Exploratory endpoint (Correlation between functional connectivity and self-reported anhedonia) | treatment day 1 and treatment day 2
  Correlation between resting state functional connectivity and self- reported anhedonia after amisulpride administration as compared to placebo in MDD patients relative to HV
Exploratory endpoint (Correlation between functional connectivity and behavioral measures) | treatment day 1 and treatment day 2
  Correlation between resting state functional connectivity and behavioral measures after amisulpride administration as compared to placebo in MDD patients relative to HV
Exploratory endpoint (Change in plasma levels of amisulpride) | treatment day 1 and treatment day 2
  Changes in plasma levels of amisulpride including correlation to changes in BOLD signal in MDD patients relative to HV
Exploratory endpoint (Change in whole brain BOLD signal) | treatment day 1 and treatment day 2
  Changes in whole brain BOLD signal after amisulpride administration as compared to placebo in MDD patients relative to HV

CONTACTS AND LOCATIONS:
Overall Officials: Christian Keicher, Dr. med., Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité Research Organisation GmbH, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carstens L, Popp M, Keicher C, Hertrampf R, Weigner D, Meiering MS, Luippold G, Sussmuth SD, Beckmann CF, Wunder A, Grimm S. Effects of a single dose of amisulpride on functional brain changes during reward- and motivation-related processing using task-based fMRI in healthy subjects and patients with major depressive disorder - study protocol for a randomized clinical trial. Trials. 2023 Nov 27;24(1):761. doi: 10.1186/s13063-023-07788-x. PMID 38012795